CLINICAL TRIAL: NCT03510494
Title: The Childhood Health, Activity, and Motor Performance School Study Denmark
Brief Title: The Svendborg-project
Acronym: CHAMPS-DK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: University College Lillebælt (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20080047
Record Dates: First submitted 2018-04-12; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Obesity, Childhood; Risk Factor, Cardiovascular; Sports Injury; Physical Activity; Motor Activity
MeSH Terms: conditions — Pediatric Obesity; Athletic Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention group receiving 270 minutes of weekly physical education Control group receiving 90 minutes of weekly physical education Intervention group physical education teachers receiving physical education courses (ATK-concept)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Trebling of weekly curricular physical education (270 minutes per week)
  Interventions: Behavioral: Augmented physical education program
- Control (No Intervention): Standard curriculum physical education (90 minutes per week)

INTERVENTIONS:
Behavioral: Augmented physical education program — Augmented physical education program
  Arms: Intervention

SUMMARY:
The main aim of this study is to describe differences in development of health and motor performance over time in relation to type of school and other background variables.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at school participating in study
* Grade 0 - 4
* written, informed consent provided by parent or legal guardian

Exclusion Criteria:

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1209 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Body weight (kilograms) | Change over 2 years
  Standardized assessments performed by trained personal using an electronic scale.
Dual-energy X-ray absorptiometry (DXA) determined bone mineral content (grams) | Change over 2 years
  Standardized assessments performed by trained personal.
Musculoskeletal problems (injuries, defined as inability to participate in sports) | Total incidence of musculoskeletal problems across 2.5 years
  Weekly short-message-service tracking of participants to determine severity, frequency and nature (acute/overuse) of injuries.
Height (centimeters) | Change over 2 years
  Standardized assessments performed by trained personal using a stadiometer.
Body-mass index (kg/m^2) | Change over 2 years
  Calculated from measured height and weight
Waist circumference (centimeters) | Change over 2 years
  Standardized assessments performed by trained personal at the level of the umbilical cord
DXA determined body fat (%) | Change over 2 years
  In subcohort only. Standardized assessments performed by trained personal.
Serum fasting insulin (IU/l) | Change over 2 years
  Standardized assessments performed by trained biomedical laboratory technicians. Fasting status affirmed verbally.
Serum fasting glucose (mmol/l) | Change over 2 years
  Standardized assessments performed by trained biomedical laboratory technicians. Fasting status affirmed verbally.
Serum fasting triglycerides (mmol/l) | Change over 2 years
  Standardized assessments performed by trained biomedical laboratory technicians. Fasting status affirmed verbally.
Serum fasting total cholesterol (mmol/l) | Change over 2 years
  Standardized assessments performed by trained biomedical laboratory technicians. Fasting status affirmed verbally.
Serum fasting low-density lipoprotein cholesterol (mmol/l) | Change over 2 years
  Standardized assessments performed by trained biomedical laboratory technicians. Fasting status affirmed verbally.
Serum fasting high-density lipoprotein cholesterol (mmol/l) | Change over 2 years
  Standardized assessments performed by trained biomedical laboratory technicians. Fasting status affirmed verbally.
Serum fasting C-reactive protein (mg/l) | Change over 2 years
  Standardized assessments performed by trained biomedical laboratory technicians. Fasting status affirmed verbally.
Homeostasis model assessment of insulin resistance (HOMA-IR) | Change over 2 years
  Calculated as fasting insulin (IU/l) x fasting glucose (mmol/l))/ 22.5
Resting systolic blood pressure (mmHg) | Change over 2 years
  Standardized assessments performed by trained personal
Resting diastolic blood pressure (mmHg) | Change over 2 years
  Standardized assessments performed by trained personal
Composite risk factor score (z-scores) | Change over 2 years
  Standardized (z-scores) values of HOMA-IR, triglycerides, cholesterol-fractions, systolic blood pressure, and cardiorespiratory fitness
Cardiorespiratory fitness (meters) | Change over 2 years
  Performance on indirect cardiorespiratory fitness test (Andersen-test). Standardized assessments performed by trained personal
Handgrip strength (kg) | Change over 2.5 years
  Maximal strength measured by a dynamometer. Standardized assessments performed by trained personal
Agility (seconds) | Change over 2.5 years
  Measured by the 50 meter short-shuttle test. Standardized assessments performed by trained personal
Backward balance (0-72 points) | Change over 2.5 years
  From the "Korperkoordinations Test fur Kinder". Standardized assessments performed by trained personal
Maximal vertical jump performance (centimeters) | Change over 2.5 years
  Standardized assessments performed by trained personal
Precision throw (0-30 points) | Change over 2.5 years
  From ''Der Allgemeiner Sportmotorischer Test fur Kinder von 6-11 Jahren''

OTHER OUTCOMES:
Physical activity determined objectively using waist-worn accelerometry. Participants will be asked to wear the monitors for at least one week. | Non-specific follow-up duration as multiple time-points are considered (follow-up at 2, 3.5 and 6.5 years)
  Physical activity outcomes include; mean count/min, light-physical activity, moderate-physical activity, vigorous-physical activity. First physical activity assessment made during year 1 of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Niels Wedderkopp, Prof, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon request from the CHAMPS Study Steering Committee due to legal and ethical restrictions. Interested parties may contact Dr Niels Wedderkopp (nwedderkopp@health.sdu.dk), and the following information will be required at the time of application: a description of how the data will be used, securely managed, and permanently deleted.

REFERENCES:
- [Background] Wedderkopp N, Jespersen E, Franz C, Klakk H, Heidemann M, Christiansen C, Moller NC, Leboeuf-Yde C. Study protocol. The Childhood Health, Activity, and Motor Performance School Study Denmark (The CHAMPS-study DK). BMC Pediatr. 2012 Aug 20;12:128. doi: 10.1186/1471-2431-12-128. PMID 22906115
- [Background] Cheron C, Leboeuf-Yde C, Le Scanff C, Jespersen E, Rexen CT, Franz C, Wedderkopp N. Leisure-time sport and overuse injuries of extremities in children age 6-13, a 2.5 years prospective cohort study: the CHAMPS-study DK. BMJ Open. 2017 Jan 13;7(1):e012606. doi: 10.1136/bmjopen-2016-012606. PMID 28087543
- [Background] Huang T, Gejl AK, Tarp J, Andersen LB, Peijs L, Bugge A. Cross-sectional associations of objectively measured physical activity with brain-derived neurotrophic factor in adolescents. Physiol Behav. 2017 Mar 15;171:87-91. doi: 10.1016/j.physbeh.2016.12.026. Epub 2016 Dec 24. PMID 28027935
- [Background] Hebert JJ, Moller NC, Andersen LB, Wedderkopp N. Organized Sport Participation Is Associated with Higher Levels of Overall Health-Related Physical Activity in Children (CHAMPS Study-DK). PLoS One. 2015 Aug 11;10(8):e0134621. doi: 10.1371/journal.pone.0134621. eCollection 2015. PMID 26262678
- [Background] Heidemann M, Holst R, Schou AJ, Klakk H, Husby S, Wedderkopp N, Molgaard C. The influence of anthropometry and body composition on children's bone health: the childhood health, activity and motor performance school (the CHAMPS) study, Denmark. Calcif Tissue Int. 2015 Feb;96(2):97-104. doi: 10.1007/s00223-014-9941-9. Epub 2014 Dec 25. PMID 25539855
- [Background] Larsen LR, Kristensen PL, Junge T, Rexen CT, Wedderkopp N. Motor Performance as Predictor of Physical Activity in Children: The CHAMPS Study-DK. Med Sci Sports Exerc. 2015 Sep;47(9):1849-56. doi: 10.1249/MSS.0000000000000604. PMID 25539477
- [Background] Klakk H, Grontved A, Moller NC, Heidemann M, Andersen LB, Wedderkopp N. Prospective association of adiposity and cardiorespiratory fitness with cardiovascular risk factors in healthy children. Scand J Med Sci Sports. 2014 Aug;24(4):e275-82. doi: 10.1111/sms.12163. Epub 2014 Jan 8. PMID 24397591
- [Result] Moller NC, Tarp J, Kamelarczyk EF, Brond JC, Klakk H, Wedderkopp N. Do extra compulsory physical education lessons mean more physically active children--findings from the childhood health, activity, and motor performance school study Denmark (The CHAMPS-study DK). Int J Behav Nutr Phys Act. 2014 Sep 24;11:121. doi: 10.1186/s12966-014-0121-0. PMID 25248973
- [Result] Heidemann M, Jespersen E, Holst R, Schou AJ, Husby S, Molgaard C, Wedderkopp N. The impact on children's bone health of a school-based physical education program and participation in leisure time sports: the Childhood Health, Activity and Motor Performance School (the CHAMPS) study, Denmark. Prev Med. 2013 Aug;57(2):87-91. doi: 10.1016/j.ypmed.2013.04.015. Epub 2013 Apr 30. PMID 23643934
- [Result] Klakk H, Chinapaw M, Heidemann M, Andersen LB, Wedderkopp N. Effect of four additional physical education lessons on body composition in children aged 8-13 years--a prospective study during two school years. BMC Pediatr. 2013 Oct 17;13:170. doi: 10.1186/1471-2431-13-170. PMID 24131778
- [Result] Klakk H, Andersen LB, Heidemann M, Moller NC, Wedderkopp N. Six physical education lessons a week can reduce cardiovascular risk in school children aged 6-13 years: a longitudinal study. Scand J Public Health. 2014 Mar;42(2):128-36. doi: 10.1177/1403494813505726. Epub 2013 Sep 20. PMID 24055828
- [Result] Jespersen E, Rexen CT, Franz C, Moller NC, Froberg K, Wedderkopp N. Musculoskeletal extremity injuries in a cohort of schoolchildren aged 6-12: a 2.5-year prospective study. Scand J Med Sci Sports. 2015 Apr;25(2):251-8. doi: 10.1111/sms.12177. Epub 2014 Jan 29. PMID 24472003
- [Derived] Wedderkopp N, Wang C, Steele R, Hebert J, Rexen C, Jespersen E, Junge T, Thomsen T, Jensen FM, Shrier I. Incidence of and Risk Factors for Lower Extremity Apophysitis in Children and Adolescents. Sports Med. 2025 Nov 3. doi: 10.1007/s40279-025-02328-w. Online ahead of print. PMID 41182572
- [Derived] Tarp J, Jespersen E, Moller NC, Klakk H, Wessner B, Wedderkopp N, Bugge A. Long-term follow-up on biological risk factors, adiposity, and cardiorespiratory fitness development in a physical education intervention: a natural experiment (CHAMPS-study DK). BMC Public Health. 2018 May 9;18(1):605. doi: 10.1186/s12889-018-5524-4. PMID 29739385